CLINICAL TRIAL: NCT05352750
Title: A Phase 1, Dose-Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SON-1010 (IL12-FHAB) in Adult Patients With Advanced Solid Tumors.
Brief Title: Phase 1 Study of SON-1010 in Adult Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sonnet BioTherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SB101
Record Dates: First submitted 2022-04-05; First posted 2022-04-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor; Soft Tissue Sarcoma Adult
Keywords: Immunotherapy; Interleukin-12; First-in-human

STUDY DESIGN:
Intervention Model Description: Dose escalation and expansion at the SON-1010 MAD with trabectedin in advanced STS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Dose Level 1 (Experimental): SON-1010 Dose Level 1
  Interventions: Biological: SON-1010
- Dose Level 2 (Experimental): SON-1010 Dose Level 2
  Interventions: Biological: SON-1010
- Dose Level 3 (Experimental): SON-1010 Dose Level 3
  Interventions: Biological: SON-1010
- Dose Level 4 (Experimental): SON-1010 Dose Level 4
  Interventions: Biological: SON-1010
- Dose Level 5 (Experimental): SON-1010 Dose Level 5
  Interventions: Biological: SON-1010
- Dose Level 6 (Experimental): SON-1010 Dose Level 6
  Interventions: Biological: SON-1010
- Expansion group using SON-1010 with trabectedin in advanced soft tissue sarcoma (Experimental): SON-1010 Dose Level 6 alternating with trabectedin
  Interventions: Biological: SON-1010

INTERVENTIONS:
Biological: SON-1010 — SON-1010 is a recombinant, single-chain, unmodified human rIL-12 joined by a flexible linker to the fully human albumin binding (FHAB) domain that "hitch-hikes" on serum albumin for transport to the tumor microenvironment.
  Other Names: IL12-FHAB

SUMMARY:
This is a Phase 1, first-in-human, open-label, adaptive-design outpatient study to assess the safety, tolerability, and PK/PD of SON-1010 administered to patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a study of SON-1010, a single-chain human Interleukin-12 (IL12) cytokine linked to a single-chain variable region (scFv) antibody fragment, known as the fully human albumin binding domain (FHAB). The albumin binding domain moiety of SON-1010 attaches to albumin in the bloodstream, resulting in significantly enhanced drug PK properties, potentially lower risk than IL12 alone, and a broader therapeutic index. The study is designed to safely establish the Recommended Phase 2 Dose (RP2D) and/or maximum tolerated dose (MTD) with up to 6 dose-escalation groups and to expand the dataset at the maximum achieved dose (MAD) in combination with trabectedin in patients with advanced soft-tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 at the time of informed consent
2. Must have histologically or cytologically verified solid epithelial or mesenchymal tumors.
3. Locally advanced or metastatic disease
4. Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST v1.1), or the modified criteria for immune-based therapeutics (termed iRECIST) as appropriate. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
5. Must have been treated with standard of care therapies for their disease and have no standard alternative treatment options that are deemed by the treating physician to offer reasonable or potentially better benefit, or not be a candidate for standard therapy for their disease due to an underlying physical condition. Note that if patients have alternative therapies available that are known to confer clinical benefit, they should be informed of these therapies during the informed consent process.
6. Must weigh >50 kg to ≤120 kg at screening (to facilitate SON-1010 dilution before dosing).
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
8. Adequate organ and bone marrow function, in the absence of growth factors, as defined by the following laboratory parameters by day -1:

   1. Hematologic: neutrophils ≥1500/μL, platelets ≥100,000/μL, lymphocytes ≥500/μL, hemoglobin ≥9 g/dL (transfusion and/or erythropoietin not permitted within 2 weeks before blood draw)
   2. Renal: estimated glomerular filtration rate ≥45 mL/min/1.73 m2 (Levey 2009)
   3. Hepatic: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x ULN or ≤5 x ULN if liver metastases; coagulation international normalized ratio (INR) and activated partial thromboplastin time (aPTT), ≤1.5 x ULN; serum total bilirubin ≤1.5 x ULN or total bilirubin ≤ULN for patients with total bilirubin >1.5 x ULN (except for elevated bilirubin secondary to Gilberts disease. Confirmation of Gilberts diagnosis requires: elevated unconjugated (indirect) bilirubin values; normal complete blood count (in previous 12 months), blood smear and reticulocyte count; normal transaminases and alkaline phosphatase in previous 12 months.
   4. Chemistry: albumin ≥3.0 g/dL at screening
9. Females of childbearing potential, <1-year postmenopause who are not permanently sterile, must have a negative serum pregnancy test (beta-human chorionic gonadotropin [β-HCG]) at baseline (unless they have had a hysterectomy), and agree to use 2 highly effective methods of birth control during the study and for 30 days after the last dose of study intervention. Females who are not of childbearing potential (have had a tubal ligation, hysterectomy, or bilateral oophorectomy, or are ≥1 year postmenopause) or have a partner who has had a vasectomy do not need to use any contraception.

   Nonchildbearing potential is defined as surgically sterile or postmenopausal (defined as 12 months of spontaneous amenorrhea). A follicle stimulating hormone (FSH) level >40 IU/L at screening will confirm postmenopausal status. If a patient is not sexually active, but becomes active, then she and her male partner must use 2 methods of adequate contraception.
10. Males and their female partners must use a highly effective method of birth control if female partner(s) is of childbearing potential and must not donate sperm during the study and for 30 days after the last dose of study intervention.
11. Willing and able to provide signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
12. Must be able to communicate well with Investigator and/or study site personnel and to comply with the requirements of the entire study.

Exclusion Criteria:

1. Known history of allergy to any component of study intervention.
2. History of severe allergic/anaphylactic reaction.
3. Infection with HIV-1 or HIV-2 or a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
4. Current active liver disease from any cause, including hepatitis A (hepatitis A virus IgM positive), hepatitis B (hepatitis B virus [HBV] surface antigen positive), or hepatitis C (hepatitis C virus [HCV] antibody positive, confirmed by HCV ribonucleic acid). Patients with HCV with undetectable virus after treatment are eligible (note: patients must have completed curative antiviral therapy at least 4 weeks before screening).
5. Pregnancy and/or lactation
6. Has received a live or live-attenuated vaccine within 28 days before the first dose of study intervention. Note: Administration of killed vaccines and COVID-19 vaccines that are not live or live-attenuated are allowed if >14 days before the first dose.
7. History of any active infection requiring systemic antibiotics, antivirals or antifungals within 14 days before the first dose of study intervention, including COVID-19 as determined by the currently recommended testing strategy for acute infection.
8. Any acute noninfectious illness not resolved by14 days before day 1.
9. History of or known or suspected autoimmune disease (exception(s): patients with vitiligo, Type I diabetes, resolved childhood atopic dermatitis, hypothyroidism, or hyperthyroidism that is clinically euthyroid at Screening are allowed). Other exceptions may be allowed following discussion with the Sponsor Medical Monitor for patients who have not received treatment for their autoimmune disorder in the past 3 years.
10. Known active central nervous system metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks before study entry and have no evidence of new or enlarging brain metastases.
11. Unresolved toxicities from prior anticancer therapy, defined as not resolved to baseline or to grade 1 by the CTCAE V 5.0 criteria (NCI 2017) except for alopecia, peripheral neuropathy, and hypothyroidism secondary to prior checkpoint inhibitor therapy if currently being treated and clinically euthyroid.
12. Receipt of any investigational agent or treatment within a period of 5 half-lives (or 28 days whichever is shorter) before the first dose of study intervention.
13. Any prior immunotherapy or treatment with checkpoint inhibitors, unless approved by the Sponsor, within a period of 5 half-lives (or 3 months, whichever is shorter) since the last dose of the therapy.
14. Use of systemic steroids >10 mg/day prednisone (or equivalent) within 14 days of enrollment, except for local (topical, nasal, or inhaled) steroid use. Limited doses of systemic steroids (eg, in patients with exacerbation of reactive airway disease) must have been completed at least 10 days before enrollment. Steroid use to prevent IV contrast allergic reaction or anaphylaxis in patients who have known contrast allergies is allowed at any time before enrollment.
15. Active known second malignancy except any of the following:

    * Adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, or Stage 0 carcinoma in situ
    * Adequately treated Stage I cancer from which the patient is currently in remission and has been in remission for ≥2 years
    * Low-risk prostate cancer with Gleason score <7 and prostate-specific antigen <10 ng/mL
    * Any other cancer from which the patient has been disease-free for ≥2 years
16. Use of biotin (ie Vitamin B7) or supplements containing biotin higher than the daily adequate intake of 30 μg (FDA 2019) (Note: patients who switch from a high dose to a dose of 30 μg/day or less are eligible).
17. Any of the following events within 6 months before baseline Day 1:

    * Myocardial infarction
    * Unstable angina
    * Unstable symptomatic ischemic heart disease
    * New York Heart Association class III or IV heart failure
    * Thromboembolic events (eg, pericardial effusion, restrictive cardiomyopathy, severe untreated valvular stenosis, or severe congenital heart disease)
18. Electrocardiogram QT interval corrected for heart rate (QTc) > 470 msec, measured by Fridericia's formula [QTcF=QT/(RR0.33)]. If the QTc is prolonged in a patient with a pacemaker or bundle branch block, the patient may be enrolled in the study if confirmed by the medical monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of SON-1010 | Through study completion, an average of 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
To establish the maximum tolerated dose (MTD) of SON-1010 | Through study completion, an average of 1 year
  Highest safe dose achieved during dose escalation

SECONDARY OUTCOMES:
Serum and urine concentrations of SON-1010 will be determined at various time points | Cycles 1 and 2 (each cycle is 28 days)
  Concentration vs time of SON-1010 will be measured using blood & urine samples taken at various time points on study
Effect of SON-1010 on Serum cytokine levels | Cycles 1 and 2 (each cycle is 28 days)
  Concentration of serum level of IL-2, IL-6, IL-10 will be measured using blood samples taken at various time points on study
Evaluation of SON-1010 immunogenicity | Cycles 1, 2 and 3 (each cycle is 21 days)
  Evaluate the immunogenicity of SON-1010 by measuring the number of patients developing anti-SON-1010 antibodies
To assess the antitumor activity of SON-1010 | Through study completion, an average of 1 year
  Objective response rate per RECIST 1.1 and iRECIST or other appropriate disease-specific response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kenney, MD, Study Director — Sonnet BioTherapeutics
Locations (1):
- Sarcoma Oncology Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No